CLINICAL TRIAL: NCT05643820
Title: Comparison of Oral Ivermectin and Permethrin 5% Lotion in Treatment of Pediculosis Capitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Combined Military Hospital Abbottabad (Other)
Responsible Party: Principal Investigator, Huma Farid, Dr. Huma Farid, Combined Military Hospital Abbottabad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMHAtd-ETH-21-Derm-22
Record Dates: First submitted 2022-11-22; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-12

CONDITIONS: Pediculosis
Keywords: ivermectin; permethrin 5% lotion
MeSH Terms: conditions — Lice Infestations | interventions — Permethrin; Ivermectin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Patients prescribed with topical 5% Permethrin lotion two applications seven days apart and applied overnight.
  Interventions: Drug: Permethrin 5% topical lotion
- group B (Active Comparator): Patients weighing greater than 15kgs prescribed with oral ivermectin 200microgram/kg two doses seven days apart
  Interventions: Drug: Ivermectin

INTERVENTIONS:
Drug: Permethrin 5% topical lotion — patients in group A prescribed with 5% topical permethrin lotion two overnight applications seven days apart
  Arms: Group A
Drug: Ivermectin — patients in group B and weighing more than 15 kgs were given oral ivermectin 200 microgram/kg two doses seven days apart
  Arms: group B

SUMMARY:
In children, pediculosis is a common ectoparasitic infestation. Infestation of head lice (Pediculus humanus capitis) causes a variety of physical symptoms, including pruritus, excoriation, cervical lymphadenopathy, and conjunctivitis1. It also has a number of negative social consequences, including parental anxiety and stigmatization of infested children2.

It is a significant public health issue that primarily affects school-aged children aged 8 to 113. In developing nations, prevalence rates of up to 40% have been reported4. The four urban areas of KPK (NWFP) reported prevalence of 36.7%5. People with a low socioeconomic background and poor hygiene are more likely to be affected6.

Pediculosis capitis has been treated using a variety of treatment modalities. They include both physician prescription and over-the-counter medications. Permethrin or ivermectin had been used topically or orally. Permethrin is a neurotoxin that is synthesized. It is a pyrethroid neurotoxic that targets voltage-sensitive Sodium ion receptors in the neurological system of the insect, triggering nerve depolarization, hyperexcitation, muscular paralysis, and, eventually, parasite death7. Ivermectin is antiparasitic medication, it is possible to treat diseases like lymphatic filariasis, and ectoparasite infestations, primarily scabies, with ivermectin because it binds to glutamate gated chloride ion receptors of invertebrates and disrupts neurotransmission8.

The rationale of this study is to study while comparing effectiveness of oral ivermectin and topical permethrin in management of pediculosis. The topical medication usage is problematic and had reported drug resistance9. There has been less regional or national research on the effectiveness of oral Ivermectin, so doctors less frequently use it in our department. Instead, the patients are treated for pediculosis capitis with topical Permethrin.

ELIGIBILITY:
Inclusion Criteria:

both genders with live detected on clinical examination and by combing wet hair with a fine toothed lice detection comb ages 8-36 years weight >15 kgs

Exclusion Criteria:

pregnancy breast feeding using any pediculicidal medication within the preceding two weeks of treatment hairstyle that may be difficult to comb

Ages: 8 Years to 36 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
comparison of oral ivermectin and 5%permethrin lotion the treatment of pediculosis capitis assessed after two applications seven days apart and reassessed at 14 days | 06 months
  treatment was considered to be effective with complete absence of symptoms i.e pruritus and the absence of live lice after combing wet hair with a fine toothed detection comb

CONTACTS AND LOCATIONS:
Overall Officials: Bushra Muzaffar, FCPS, Principal Investigator — Combined Military Hospital Abbottabad
Locations (1):
- CMH, Abbottabad, KPK, Pakistan